CLINICAL TRIAL: NCT00567918
Title: Phase III, Long-Term, Open-Label, Extension Study of 0.1% Tacrolimus(FK506) Ophthalmic Suspension in Patients
Brief Title: Phase III, Long-Term, Open-Label, Extension Study of 0.1% Tacrolimus(FK506) Ophthalmic Suspension in Patients With Vernal Keratoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ-506D-AC10
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: Keratoconjunctivitis; Conjunctivitis
Keywords: Keratoconjunctivitis; Vernal keratoconjunctivitis; FK506; Tacrolimus
MeSH Terms: conditions — Keratoconjunctivitis; Conjunctivitis; Conjunctivitis, Allergic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): FK506 ophthalmic suspension
  Interventions: Drug: FK506

INTERVENTIONS:
Drug: FK506 — Ophthalmic suspension
  Other Names: tacrolimus

SUMMARY:
To investigate the long-term efficacy and safety of FK506 ophthalmic suspension in patients with vernal keratoconjunctivitis

DETAILED DESCRIPTION:
To give a chance of continuous use of 0.1% FK506 ophthalmic suspension to patients with vernal keratoconjunctivitis who were enrolled in the FJ-506D-AC09 study, long-term safety and efficacy were evaluated. Primary efficacy endpoint was the mean change from the baseline (before the treatment) in total score for objective clinical signs.

ELIGIBILITY:
Inclusion Criteria:

* Vernal keratoconjunctivitis patients who were enrolled in the FJ-506D-AC09 study
* Patients who wish to receive continuous administration of FK506 ophthalmic suspension

Exclusion Criteria:

* Subjects who needed prohibited concomitant therapy at the initiation of the study
* Subjects who needed to wear contact lenses during treatment period on a testing eye
* Subjects with complicating an eye infection

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Safety | length of study

SECONDARY OUTCOMES:
The mean change from the baseline (before the treatment) in total score for objective clinical signs | length of study
Mean change from the baseline in score for objective clinical signs and the score for each objective clinical sign | Length of study
Subjective symptom score (Visual Analog Scale) | Length of study
The improvement rate | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Ehime
  - Hokkaido
  - Kagoshima
  - Kochi
  - Miyazaki
  - Osaka
  - Tochigi
  - Tokyo